CLINICAL TRIAL: NCT06132841
Title: A Phase I Randomized, Single-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD6234 Following Repeat Dose Administration in Participants With Overweight or Obesity
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD6234 After Repeat Dose Administration in Participants Who Are Overweight or Obese
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: D8750C00002
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Healthy Participants
Keywords: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants will receive repeated doses of AZD6234 or placebo via SC injection
  Interventions: Drug: AZD6234; Drug: Placebo
- Cohort 2 (Experimental): Participants will receive repeated doses of AZD6234 or placebo via SC injection
  Interventions: Drug: AZD6234; Drug: Placebo
- Cohort 3 (Experimental): Japanese participants will receive repeated doses of AZD6234 or placebo via SC injection
  Interventions: Drug: AZD6234; Drug: Placebo
- Cohort 4 (Experimental): Japanese participants with childbearing potential will receive repeated doses of AZD6234 or placebo via SC injection.
  Interventions: Drug: AZD6234; Drug: Placebo

INTERVENTIONS:
Drug: AZD6234 — Participants will receive repeated doses of AZD6234 as a solution via SC
Drug: Placebo — Participants will receive matching volumes of the placebo as a solution via SC

SUMMARY:
A study in healthy male and female participants of non-childbearing and childbearing potential who have overweight or obesity

DETAILED DESCRIPTION:
The study will comprise of:

* A Screening Period of maximum 32 days (from Day -35 to Day -3).
* A Treatment Period of 6 weeks (Cohort 1), 12 weeks (Cohort 2 and 3) and 26 weeks (Cohort 4) during which the participants will receive the study drug during residency at clinical unit.
* A Follow-up Visit after the last dose of study drug.

This study with repeated dosing of AZD6234 consists of 4 cohorts. For cohorts 1,2 and 3, eligible participants will be randomized to AZD6234 and placebo in a 3:1 ratio. For Cohort 4, eligible participants will be randomized in a 4:1:4:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating and must be of non-childbearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.
* Have a BMI between 25 and 40 kg/m2 inclusive (at the time of screening) and weigh at least 60 kg.
* Participant must have an evaluable, pre-randomization MRI, as confirmed by the core laboratory review (Cohort 4 only).
* Cohort 4 only: Females of childbearing potential who use adequate protection (oral contraceptives are not permitted).

Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal STT wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
* Known or suspected history of drug abuse, smoking, alcohol abuse or cotinine at screening.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD6234.
* Has received prescription or non-prescription medication for weight loss within the last 3 months.
* Self-reported weight change of > 5 kg in the last 3 months prior to screening.
* Previous or planned (within study period) bariatric surgery or fitting of a weight loss device (eg, gastric balloon or duodenal barrier).
* Participants who follow vegan diet or have medical dietary restrictions.
* Participants who cannot communicate reliably with the Investigator.
* Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Contra-indication to MRI: such as participants with pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or other conditions that would preclude proximity to a strong magnetic field; participants with history of extreme claustrophobia or participant cannot fit inside the MRI scanner cavity (Cohort 4 only).

Ages: 18 Years to 142 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious Adverse Events(SAE) | From Screening (Day -35 to Day -3) to Day 78 (Cohort 1) or to Day 120 (Cohort 2 and 3) or to Day 225 (Cohort 4)
  The safety and tolerability of repeated subcutaneous (SC) doses of AZD6234 compared to placebo will be assessed.

SECONDARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | From Day 1 to Day 78 (Cohort 1) or to Day 120 (Cohort 2 and 3) or to Day 225 (Cohort 4)
  The pharmacokinetics (PK) of AZD6234 following repeated SC doses of AZD6234 will be assessed.
Area under the plasma concentration-time (AUClast) | From Day 1 to Day 78 (Cohort 1) or to Day 120 (Cohort 2 and 3) or to Day 225 (Cohort 4)
  The PK of AZD6234 following repeated SC doses of AZD6234 will be assessed.
Area under plasma concentration-time curve from zero to infinity (AUCinf) | From Day 1 to Day 78 (Cohort 1) or to Day 120 (Cohort 2 and 3) or Day 225 (Cohort 4)
  The PK of AZD6234 following repeated SC doses of AZD6234 will be assessed.
Area under concentration time curve in the dosing interval (AUCtau) | From Day 1 to Day 78 (Cohort 1) or to Day 120 (Cohort 2 and 3) or to Day 225 (Cohort 4)
  The PK of AZD6234 following repeated SC doses of AZD6234 will be assessed.
Change from baseline in body weight of participants | From baseline (Day -1) to Day 43 (Cohort 1) or to Day 85 (Cohort 2 and 3) or to Day 183 (Cohort 4)
  The effects of AZD6234 on body weight change from baseline with and without placebo correction will be assessed.
Change from baseline in Body Mass Index (BMI) of participants | From baseline (Day -1) to Day 43 (Cohort 1) or to Day 85 (Cohort 2 and 3) or to Day 183 (Cohort 4)
  The effects of AZD6234 on body weight change from baseline with and without placebo correction will be assessed.
Percentage change from baseline in fasting insulin | From baseline (Day -1) to Day 43 (Cohort 1) or to Day 85 (Cohort 2 and 3) or to Day 183 (Cohort 4)
  The effects of AZD6234 compared to placebo on fasting insulin will be assessed.
Change from baseline in absolute level of fasting insulin of participants | From baseline (Day -1) to Day 43 (Cohort 1) or to Day 85 (Cohort 2 and 3) or to Day 183 (Cohort 4)
  The effects of AZD6234 compared to placebo on fasting insulin will be assessed.
Prevalence of anti-drug antibodies (ADAs) to AZD6234 | Day 1, 15, 36, and 78 (Cohort 1); Day 1, 15, 29, 43, 78 and 120 (Cohort 2 and 3) or to Day 183 (Cohort 4)
  The immunogenicity of AZD6234 following repeated SC doses of AZD6234 will be assessed.
Incidence of ADAs to AZD6234 | Day 1, 15, 36, and 78 (Cohort 1); Day 1, 15, 29, 43, 78 and 120 (Cohort 2 and 3) to Day 183 (Cohort 4)
  The immunogenicity of AZD6234 following repeated SC doses of AZD6234 will be assessed.
ADA titer | Day 1, 15, 36, and 78 (Cohort 1); Day 1, 15, 29, 43, 78 and 120 (Cohort 2 and 3) or to Day 183 (Cohort 4)
  The immunogenicity of AZD6234 following repeated SC doses of AZD6234 will be assessed.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Brooklyn, Maryland
- Research Site, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/